CLINICAL TRIAL: NCT00530452
Title: Double-Blind, Placebo Controlled Phase II Repeat Dose Study of the Safety and Efficacy of Three Parallel Loading and Maintenance Dose Regimens of CG100649 Versus Placebo for the Treatment of Primary Osteoarthritis in Male Subjects
Brief Title: Phase II Study of CG100649 for Primary Osteoarthritis in Male Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CrystalGenomics, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: William K. Schmidt, PhD, CrystalGenomics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG100649-2-01; EudraCT number: 2007-001197-93
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: COX-2; carbonic anhydrase; osteoarthritis; anti-inflammatory; Cyclooxygenase Inhibitors
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis | interventions — CG100649; Talc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): 2.0 mg (loading dose, Day 0) followed by 0.3 mg/day (Days 1-20)
  Interventions: Drug: CG100649
- B (Experimental): 4.0 mg (loading dose, Day 0) followed by 0.6 mg/day (Days 1-20)
  Interventions: Drug: CG100649
- C (Experimental): 8.0 mg (loading dose, Day 0) followed by 1.2 mg/day (Days 1-20)
  Interventions: Drug: CG100649
- D (Placebo Comparator): Placebo (identical number of capsules to active drug groups) (Days 0-20)
  Interventions: Drug: Silicified microcrystalline cellulose + talc

INTERVENTIONS:
Drug: CG100649 — Dual-acting COX-2 inhibitor & carbonic anhydrase inhibitor in gelatin capsules. Oral loading doses (2, 4, or 8 mg vs. placebo) followed by daily oral maintenance doses (0.3, 0.6, or 1.2 mg vs. placebo) for 20 days (total 21 days therapy).
  Arms: A; B; C
Drug: Silicified microcrystalline cellulose + talc — Gelatin capsules containing cellulose/talc matched for weight and color to experimental medication. Placebo administered orally 1x/day.
  Arms: D

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of 3 loading and maintenance dose levels of CG100649 administered for 21 days in the treatment of osteoarthritis pain.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled study. Subjects will discontinue current medications 5-14 days prior to randomization. Paracetamol (acetaminophen; ≤2 gm/day) may be used for breakthrough pain. Other NSAIDs, COX-2 inhibitors, opioids, and corticosteroids may not be used at any time during this study. Only subjects recording average DPI of 4 to 8 on a 0-10 numerical rating scale for at least 3 days, and no greater than 9 for more than 1 day, during the last 5 days of the washout period and meeting all other inclusion criteria will be randomized into the study.

Subjects meeting screening criteria will be randomized to receive 21 days dosing of an active dose of CG100649 or placebo.

Antiarthritic efficacy will be evaluated by changes in the Western Ontario and McMaster Universities (WOMAC) OA index completed on Day 0 (Baseline) and on Days 7, 14, 21, 28, and 35. DPI and functional interference (BPI scales) will be evaluated by subject diary during the screening period and on all study days through Day 35. Pain Relief will be evaluated on Days 7, 14, 21, 28, and 35.

ELIGIBILITY:
Inclusion Criteria:

1. Males, age 18-75 years old;
2. BMI 19-35 kg/m2;
3. Good health;
4. Systolic BP 90-140 mmHg, diastolic BP 50-90 mmHg, resting HR 45-90 bpm without medication;
5. Clinical chemistry profile within 2x normal range without medication;
6. Urinalysis including urinary creatinine within 2x normal limits;
7. OA confirmed by radiographs obtained within the past 20 years and diagnosed according to ACR guidelines; subjects must qualify as ACR global functional status I, II, or III (excluding IV) and Kellgren-Lawrence grade 1, 2 or 3 (excluding grades 0 and 4);
8. Subjects must have had chronic pain for ≥3 months from OA;
9. Subjects must have been receiving stable oral doses of NSAIDs or COX-2 inhibitors at least 3 days per week for one month or longer;
10. Subjects may take paracetamol ≤2g/day) for breakthrough pain;
11. During the washout period, the average daily pain intensity (DPI) score must be between 4 and 8 on a 0-10 numerical rating scale for at least 3 days, and no greater than 9 for more than 1 day, in the last 5 days prior to randomization per Baseline pain diary;
12. Subjects must be able to read, understand and follow the study instructions;
13. Subjects and their sexual partners must agree to use double barrier contraception during the study period and for 2 months afterward.

Exclusion Criteria:

1. Use of any analgesics except the study medication or paracetamol;
2. Presence or history of peripheral edema within the past 5 years;
3. History of congestive heart failure;
4. Use of chemotherapy agents or history of cancer within five years prior to the screening visit;
5. History of bacterial or viral infection requiring treatment with antibiotics, antivirals, or anti-retrovirals within 3 months of study;
6. Use of drugs which are P450 3A4 inducers or inhibitors within the past 30 days;
7. Use of prescribed systemic or topical medications or any dietary aids or foods that are known to modulate drug metabolizing enzymes within 14 days of dose administration;
8. Difficulty in swallowing oral medications;
9. Subjects with gout, pseudogout, inflammatory arthritis, Paget's disease of bone, chronic pain syndrome, fibromyalgia, or another major joint disease;
10. Subjects requiring knee or hip arthroplasty within 2 months of screening or anticipating any need for a surgical procedure on the index joint during the study;
11. Subjects who have had surgery on the affected joint within one year prior to the study and subjects with a prosthesis at the index joint;
12. Use of systemic corticosteroids within 2 months of screening, or intra-articular viscosupplementation within the past 6 months;
13. History of seizure disorder;
14. Use of antidepressants or anticonvulsants for any reason including for chronic pain within 2 months of screening;
15. Serious psychosocial co-morbidities;
16. Cognitive or psychiatric disorders, or daytime use of medications that could diminish compliance with study procedures, including maintenance of a daily pain and symptom diary and accurate dosing of study medication;
17. Use of anticoagulants within 2 weeks of screening;
18. Use of any medications that will affect pain perception;
19. History of drug or alcohol abuse within one year prior to screening;
20. Use of any other investigational drug within 1 month prior to randomization;
21. Active gastrointestinal, renal, hepatic, or coagulant disorder within 1 month prior to randomization;
22. Esophageal or gastroduodenal ulceration within 1 month prior to randomization;
23. Hypersensitivity to NSAIDs, sulfonamides, COX-2 inhibitors, or carbonic anhydrase inhibitors;
24. History of nasal polyps, bronchospasm or urticaria;
25. Known allergy or hypersensitivity to sulfa drugs;
26. Family history of significant cardiac disease;
27. Occult blood in stool.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the change in the sum of the WOMAC OA index at Day 21 vs. Baseline (Day 0). The primary analysis will be via repeated measures using mixed effects ANOVA with baseline and subject as random variables. | 21 days

SECONDARY OUTCOMES:
Change in av. Daily Pain Intensity (DPI) during last 7 days & entire 21 days); • Change in worst DPI (last 7 days; entire 21 days); • Change in WOMAC OA index on Days 7, 14, 28, and 35 vs. baseline; • Subject's Global Assessment • Safety | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — CrystalGenomics, Inc.
Locations (1):
- Orthopaedische Praxis, Bad Dürrheim, Baden-Wurttemberg, Germany